CLINICAL TRIAL: NCT00346268
Title: Randomized, Double-Blind Study Of The Morphine-Sparing Efficacy And Safety Of Parecoxib Sodium 40 Mg IV Followed By 20 Mg IV Every 12 Hours In The Treatment Of Pain Following Radical Prostatectomy
Brief Title: Morphine-Sparing Efficacy Of Parecoxib In Pain Treatment After Radical Prostatectomy
Acronym: PROSTATECTOMY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3481066
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Results first posted 2011-10-28 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; parecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine plus Parecoxib (Active Comparator)
  Interventions: Drug: Morphine, Parecoxib
- Morphine and Placebo (Active Comparator)
  Interventions: Drug: Morphine, Placebo

INTERVENTIONS:
Drug: Morphine, Parecoxib — Parecoxib 40 milligrams (mg) administered intravenously immediately post surgery, followed 20 mg every 12 hours until 48 hours post surgery, total 5 doses. Participants also received Patient-Controlled Analgesia (PCA) 1 mg per dose, maximum 40 mg/4 hours, and if necessary, bolus (2 to 5 mg) before or after enabled PCA.
  Arms: Morphine plus Parecoxib
Drug: Morphine, Placebo — Matching placebo administered intravenously immediately post surgery and every 12 hours until 48 hours post surgery, total 5 doses. Participants also received PCA (1 mg per dose, maximum 40 mg/4 hours, and if necessary, bolus (2 to 5 mg) before or after enabled PCA
  Arms: Morphine and Placebo

SUMMARY:
The primary objective of this study is to demonstrate the opioid-sparing efficacy of parecoxib 40 mg intravenously given as a loading dose followed by 20 mg intravenously in the 24 hours after the end of surgery.

DETAILED DESCRIPTION:
The study was terminated due to lack of recruitment due to competing alternative operation methods on 13September 2010. The decision to terminate the trial was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* The patient's ASA physical status is 1 or 2 and he has a low risk (i.e.,<10%) of developing an acute coronary event within the next 10 years according to the PROCAM risk assessment calculator.
* The patient is scheduled to undergo routine radical prostatectomy performed under a standardized regimen of general anesthesia, and is expected to experience moderate to severe postsurgical pain in the absence of postoperative analgesia.

Exclusion Criteria:

* The patient has a history of uncontrolled chronic disease or a concurrent clinically significant illness or medical condition such as a diagnosed chronic pain condition, which, in the Investigator's opinion, would contraindicate study participation or confound interpretation of the results
* The patient has a history or current presence of congestive heart failure (NYHA II-IV), established ischaemic heart disease, peripheral arterial disease and / or cerebrovascular disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Germany (4):
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Reutlingen

REFERENCES:
- [Derived] Dirkmann D, Groeben H, Farhan H, Stahl DL, Eikermann M. Effects of parecoxib on analgesia benefit and blood loss following open prostatectomy: a multicentre randomized trial. BMC Anesthesiol. 2015 Mar 9;15:31. doi: 10.1186/s12871-015-0015-y. eCollection 2015. PMID 25767411
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3481066&StudyName=Morphine-Sparing%20Efficacy%20Of%20Parecoxib%20In%20Pain%20Treatment%20After%20Radical%20Prostatectomy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was terminated prematurely due to slow recruitment.
Groups:
- Parecoxib and Morphine: Parecoxib 40 milligrams (mg) administered intravenously immediately post surgery, followed 20 mg every 12 hours until 48 hours post surgery, total 5 doses. Participants also received Patient-Controlled Analgesia (PCA) 1 mg per dose, maximum 40 mg/4 hours, and if necessary, bolus (2 to 5 mg) before or after enabled PCA.
- Placebo and Morphine: Matching placebo administered intravenously immediately post surgery and every 12 hours until 48 hours post surgery, total 5 doses. Participants also received PCA (1 mg per dose, maximum 40 mg/4 hours, and if necessary, bolus (2 to 5 mg) before or after enabled PCA.
Period: Overall Study
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Started | 52 | 53
Completed | 50 | 50
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Participant refused | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parecoxib and Morphine | Placebo and Morphine | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Customized [Number; unit: participants]
  < 45 years | 0 | 0 | 0
  Between 45 and 59 years | 14 | 13 | 27
  Between 60 and 74 years | 36 | 38 | 74
  >= 75 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 52 | 53 | 105

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Amount of Morphine Administered in the First 24 Hours Following Surgery
Description: Total cumulative amount of morphine administered (PCA and/or bolus) in the first 24 hours after the application of the last surgical stitch after prostatectomy.
Time Frame: 24 hours post surgery
Population: Full Analysis Set Population (FAS): participants who were randomized to treatment
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 52 | 53
mL | 28.84 (16.16) | 36.40 (19.99)
Statistical Analysis 1: Comparison: Parecoxib and Morphine vs Placebo and Morphine; Test type: Superiority or Other; p = 0.035, ANOVA — Adjusted for treatment group and center; least square (LS) mean difference (net) = -7.58, 95% CI 2-sided [-14.63 to -0.53], Standard Error of Mean 3.55

2. Secondary Outcome: Cumulative Amount of Morphine Administered in the First 48 Hours Following Surgery
Description: Total cumulative amount of morphine administered (PCA and/or bolus) in the first 48 hours after the application of the last surgical stitch after prostatectomy.
Time Frame: 48 hours post surgery
Population: FAS
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 52 | 53
mL | 42.13 (25.02) | 57.03 (28.07)
Statistical Analysis 1: Comparison: Parecoxib and Morphine vs Placebo and Morphine; Test type: Superiority or Other; p = 0.004, ANOVA — Adjusted for treatment group and center; least square (LS) mean difference (net) = -15.16, 95% CI 2-sided [-25.47 to -4.85], Standard Error of Mean 5.20

3. Secondary Outcome: Time to Last Administration of Morphine
Description: Time from last surgical stitch after prostatectomy to last administration of morphine (PCA and/or bolus).
Time Frame: baseline (end of surgery) to 48 hours post surgery
Population: FAS; Number of participants analyzed (N)=participants with evaluable data
Measure: Median (Full Range); unit: hours
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 48 | 49
hours | 46.5 [1.9 to 123.7] | 46.5 [21.8 to 90.3]
Statistical Analysis 1: Comparison: Parecoxib and Morphine vs Placebo and Morphine; Test type: Superiority or Other; p = 0.257, Log Rank; Stratified by center

4. Secondary Outcome: Amount of Blood Loss
Description: Calculated as: ([Hb g/dL]pra + RBCUduring48)-[Hb g/dL]at 48, where [Hb g/dL]pra=blood hemoglobin concentration preoperatively in grams per deciliter (g/dL), [Hb g/dL]at 48=blood hemoglobin concentration 48 hours after skin closure, and RBCUduring48=number of red blood cell units (RBCU) substituted during and after prostatectomy until 48 hours after skin closure.
Time Frame: 48 hours post surgery
Population: FAS
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 52 | 53
g/dL | 4.34 (1.40) | 4.41 (2.12)
Statistical Analysis 1: Comparison: Parecoxib and Morphine vs Placebo and Morphine; Test type: Superiority or Other; p = 0.810, ANCOVA — Adjusted for treatment group and center; Covariates:Total RBCUs and RBCUs substituted during surgery, baseline hemoglobin, swab and lavage weights, intraoperative blood loss fluid volume; LS mean difference (net) = -0.07, 95% CI 2-sided [-0.68 to 0.53], Standard Error of Mean 0.30

5. Secondary Outcome: Number of Participants With Blood Loss Requiring Red Blood Cell (RBC) Transfused Units
Time Frame: 48 hours post surgery
Population: FAS
Measure: Number; unit: participants
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 52 | 53
participants
  1 RBC transfused unit | 1 | 1
  2 RBC transfused units | 4 | 1

6. Secondary Outcome: Pain Intensity Score
Description: Pain intensity assessed immediately prior and 30 minutes after administration (admin) of study medication, participants categorized their pain intensity at rest and at movement on 0-4 numeric rating scale (NRS):0 (minimum intensity) to 4 (maximum intensity).
  Movement defined as sitting up from a lying into a sitting position in bed.
Time Frame: 12, 24, 36, and 48 hours post surgery
Population: FAS; N=participants with evaluable data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 51 | 52
scores on a scale
  At rest, prior to admin, 12 hours post surgery | 1.31 (0.76) | 1.69 (0.95)
  At rest, post admin, 12 hours post surgery | 0.53 (0.67) | 0.79 (0.78)
  At movement, prior to admin, 12 hours post surgery | 2.12 (0.86) | 2.63 (0.95)
  At movement, post admin, 12 hours post surgery | 1.16 (0.88) | 1.58 (1.02)
  At rest, prior to admin, 24 hours post surgery | 1.00 (0.82) | 1.44 (0.94)
  At rest, post admin, 24 hours post surgery | 0.53 (0.76) | 0.67 (0.73)
  At movement, prior to admin, 24 hours post surgery | 2.12 (0.86) | 2.63 (0.77)
  At movement, post admin, 24 hours post surgery | 1.45 (1.05) | 1.90 (0.96)
  At rest, prior to admin, 36 hours post surgery | 0.86 (0.94) | 1.04 (0.87)
  At rest, post admin, 36 hours post surgery | 0.45 (0.61) | 0.59 (0.73)
  At movement, prior to admin, 36 hours post surgery | 1.59 (0.98) | 2.12 (1.03)
  At movement, post admin, 36 hours post surgery | 1.04 (0.89) | 1.51 (0.92)
  At rest, prior to admin, 48 hours post surgery | 0.67 (1.07) | 0.82 (0.97)
  At rest, post admin, 48 hours post surgery | 0.29 (0.54) | 0.29 (0.58)
  At movement, prior to admin, 48 hours post surgery | 1.47 (1.16) | 2.31 (0.97)
  At movement, post admin, 48 hours post surgery | 0.88 (0.86) | 1.41 (0.98)
Statistical Analysis 1: Comparison: Parecoxib and Morphine vs Placebo and Morphine; The difference in pain at rest prior to administration and pain at rest post administration compared between treatments at 48 hours post surgery; Test type: Superiority or Other; p = 0.070, ANOVA; Least squares mean difference (net) = 0.17, 95% CI 2-sided [-0.01 to 0.35], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Parecoxib and Morphine vs Placebo and Morphine; The difference in pain at movement prior to administration and pain at movement post administration compared between treatments at 48 hours post surgery; Test type: Superiority or Other; p = 0.074, ANOVA; LS Mean Difference (net) = 0.16, 95% CI 2-sided [-0.02 to 0.33], Standard Error of Mean 0.09

7. Secondary Outcome: Modified Brief Pain Inventory-Short Form (mBPI-sf): Pain Severity Composite Score
Description: mBPI-sf: participant-rated 11-point Likert rating scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine). Pain severity index=the mean of item scores 2 to 5 (pain at its worst in past 24 hours, pain at its least in past 24 hours, average pain level, and pain right now).
Time Frame: 24 and 48 hours post surgery
Population: FAS; N=participants with evaluable data; n=participants with evaluable for specified category; for analyses, missing values imputed using Last-Observation-Carried-Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 49 | 50
scores on a scale
  24 hours post surgery (n=49, 50) | 2.08 (1.17) | 2.78 (1.06)
  48 hours post surgery (n=43, 48) | 1.60 (1.26) | 2.31 (1.17)
Statistical Analysis 1: Comparison: Parecoxib and Morphine vs Placebo and Morphine; 24 hours post surgery; Test type: Superiority or Other; p = 0.002, ANOVA — Adjusted for treatment group and center; LS mean difference (net) = -0.71, 95% CI 2-sided [-1.16 to -0.26], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Parecoxib and Morphine vs Placebo and Morphine; 48 hours post surgery; Test type: Superiority or Other; p = 0.004, ANOVA — Adjusted for treatment group and center; LS mean difference (net) = -0.73, 95% CI 2-sided [-1.22 to -0.23], Standard Error of Mean 0.25

8. Secondary Outcome: Modified Brief Pain Inventory-Short Form (mBPI-sf): Pain Interference Composite Score
Description: mBPI-sf: participant-rated 11-point Likert rating scale ranging from 0 (does not interfere) to 10 (completely interferes) with functional activities (general activity, mood, walking ability, relations with other people, sleep, coughing, deep breathing, and concentration) in past 24 hours.
Time Frame: 24 and 48 hours post surgery
Population: FAS; N=participants with evaluable data; n=participants with evaluable data for specified category; for analyses, missing values imputed using LOCF method.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 49 | 50
scores on a scale
  24 hours post surgery (n=49, 50) | 1.16 (1.21) | 2.32 (1.78)
  48 hours post surgery (n=43, 48) | 1.00 (1.41) | 1.79 (1.50)
Statistical Analysis 1: Comparison: Parecoxib and Morphine vs Placebo and Morphine; 24 hours post surgery; Test type: Superiority or Other; p = 0.001, ANOVA — Adjusted for treatment group and center; LS mean difference (net) = -1.16, 95% CI 2-sided [-1.77 to -0.56], Standard Error of Mean 0.30
Statistical Analysis 2: Comparison: Parecoxib and Morphine vs Placebo and Morphine; 48 hours post surgery; Test type: Superiority or Other; p = 0.006, ANOVA — Adjusted for treatment group and center; LS mean difference (net) = -0.83, 95% CI 2-sided [-1.41 to -0.24], Standard Error of Mean 0.30

9. Secondary Outcome: Opiate Related Symptom Distress Scale (OR-SDS) Questionnaire: Overall Composite Score
Description: Participant-rated scale assessed 10 common opiate related symptoms by 3 ordinal measures: frequency (1 to 4 scale: rarely to almost constantly), severity (1 to 4 scale: slight to very severe) and bothersomeness (1 to 5 scale: not at all to very much). Frequency and severity items assigned numeric scores 1 to 4. Bothersomeness items scaled in order to assign numeric scores 0.8 to 4.0 (not at all scored=0.8, a little bit=1.6, somewhat=2.4, quite a bit=3.2, and very much=4.0). Overall composite score=mean of each 10 individual mean symptoms' OR-SDS scores; ranged from 1 to 4.
Time Frame: 24 and 48 hours post surgery
Population: FAS; N=participants with evaluable data.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 51 | 52
scores on scale
  24 hours post surgery | 0.50 (0.35) | 0.55 (0.39)
  48 hours post surgery | 0.26 (0.28) | 0.34 (0.34)

10. Other Pre Specified Outcome: Number of Participants With Rating of Global Evaluation of Study Medication
Description: Participants asked, "How would you rate the study medication you received for pain since your surgery?" choices included: Poor, Fair, Good, and Excellent.
Time Frame: 48 hours post surgery
Population: FAS; N=participants with evaluable data.
Measure: Number; unit: participants
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 50 | 50
participants
  Poor | 1 | 3
  Fair | 3 | 5
  Good | 19 | 31
  Excellent | 27 | 11

11. Other Pre Specified Outcome: Number of Participants With Health Care Resource Utilization (HCRU)
Description: Supervising physician or nurse answered question in the presence of participant, "In the last 24 hours, did the participant receive any unscheduled consultation from any of the following specialist: anesthesiologist, surgeon, nurse or other specialist".
Time Frame: 24 and 48 hours post surgery
Population: Data not analyzed due to study termination.
Measure: Number; unit: participants
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Overall Analgesic Benefit Score (OABS)
Description: Participants' rating of global assessment of analgesic experience. OABS comprised of scores for symptoms (vomiting, itching, sweating, freezing, and dizziness) and patient satisfaction; Participants asked how much did symptoms distress and bother them during the last 24 hours; Participants asked how satisfied they have been with treatment of pain during last 24 hours. Each symptom and satisfaction question scored from 0 (not at all) to 4 (very much so). Total possible score=0 to 24.
Time Frame: 24 and 48 hours post surgery
Population: Data not analyzed due to study termination.
Measure: Number; unit: scores on a scale
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Hemoglobin Concentration
Time Frame: 24 hours post surgery
Population: Data not analyzed due to study termination.
Measure: Number; unit: g/dL
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Total Amount of Postoperative Drainage Fluid
Description: After removal of the prostate and placement of the urine catheter, at least one easy-flow drainage was placed in the perivesical space. Drainage fluid (a mixture with a variable combination of blood and urine) was measured.
Time Frame: 24 hours post surgery
Population: Data not analyzed due to study termination.
Measure: Number; unit: mL
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Parecoxib and Morphine | Placebo and Morphine
Serious Adverse Events (participants affected / at risk) | 12/52 | 5/53
Other Adverse Events (participants affected / at risk) | 35/52 | 38/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Parecoxib and Morphine (N=52) | Placebo and Morphine (N=53)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Infected lymphocele (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Lymphatic fistula (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 4 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Parecoxib and Morphine (N=52) | Placebo and Morphine (N=53)
Anaemia (Blood and lymphatic system disorders) | 6 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 4 | 8
Flatulence (Gastrointestinal disorders) | 6 | 10
Nausea (Gastrointestinal disorders) | 12 | 16
Vomiting (Gastrointestinal disorders) | 9 | 4
Pyrexia (General disorders) | 1 | 4
Urinary tract infection (Infections and infestations) | 6 | 7
Insomnia (Psychiatric disorders) | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hypertension (Vascular disorders) | 6 | 4

LIMITATIONS AND CAVEATS:
This study was terminated prematurely due to slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.